CLINICAL TRIAL: NCT03270579
Title: An Open-Label Study to Investigate the Regional Brain Kinetics of the Positron Emission Tomography Ligand [18F]JNJ-64511070
Brief Title: A Study to Investigate the Regional Brain Kinetics of the Positron Emission Tomography Ligand [18F]JNJ-64511070
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108379; 2017-002262-47 (EudraCT Number); 64140284EDI1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: [18F]JNJ-64511070 (Experimental): Participants will receive an intravenous (IV) bolus injection of [18F]JNJ-64511070 at a dose of 185 megaBecquerel (MBq) on Day 1 of Part A to investigate the total body biodistribution and measure the radiation dosimetry of [18F]JNJ-64511070.
  Interventions: Drug: [18F]JNJ-64511070
- Part B: [18F]JNJ-64511070 (Experimental): Participants will receive an IV bolus injection of [18F]JNJ-64511070 at a dose of 185 MBq on Day 1 of Part B to measure the uptake, binding, distribution, and washout of [18F]JNJ-64511070 and to model the tissue specific kinetics of [18F]JNJ-64511070 in the human brain with the appropriate arterial IF.
  Interventions: Drug: [18F]JNJ-64511070

INTERVENTIONS:
Drug: [18F]JNJ-64511070 — An IV injection of 185 MBq [18F]JNJ-64511070 will be administered.

SUMMARY:
The main purpose of the study is to measure the whole-body distribution and radiation dosimetry of [18F]JNJ-64511070 in healthy male participants by positron emission tomography (PET) (Part A); and to measure the uptake, binding, distribution, and washout of [18F]JNJ-64511070 in the brain of healthy male participants by PET and to model tissue specific kinetics of [18F]JNJ-64511070 with the appropriate arterial input function (IF) (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) inclusive
* Nonsmoker (not smoked for 3 months prior to screening)
* Is willing to allow the investigators to place an arterial catheter in the radial artery and is assessed via physical examination (Allen test) to be a good candidate for arterial catheter placement (Part B only)
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, a man: a) who is sexually active with a woman of childbearing potential and has not had vasectomy must agree to use a condom and their female partner should also use a highly effective method of birth control for at least the same duration; b) who is sexually active with a woman who is pregnant must use a condom; c) must agree not to donate sperm
* Participants must have signed an informed consent document indicating that they understand the purpose of, and procedures required for,the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Exposed to greater than (>) 1 milliSievert (mSv) of ionizing radiation participating as a participant in research studies in the 12 months before the start of enrolment in this study
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or admission. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to both the investigator are acceptable
* Clinically significant abnormal physical and neurological examination, vital signs or 12-lead electrocardiogram (ECG) at screening or admission
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, coagulation abnormalities, or other conditions that the Investigator considers should exclude the participant and preclude their ability to participate in study procedures. Participants with a history significant liver or renal disease, or difficulty in urination, which could affect the metabolism and elimination of the radiotracer or radiometabolites should be excluded. Participants with a history of epilepsy or fits or unexplained black-outs or loss of consciousness should also be excluded
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibodies or human immunodeficiency (HIV) antibodies unless the participant has been successfully treated for HCV or HIV. In such cases, the response should be confirmed with RNA testing for the relevant pathogen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Part A: Effective Radiation Dose Following Injection of [18F]JNJ-64511070 | Up to 5 hours on Day 1
  The tissue radioactivity will be measured per organ for up to 5 hours after injection of up to 185 megaBecquerel (MBq) of [18F]JNJ-64511070 and corrected for attenuation by computed tomography (CT) transmission scans using positron emission tomography (PET) /CT. These measurements will be used to estimate effective radiation dose per organ and total body.
Part B: Total and Regional Brain Compartmental Kinetics for Volume of Distribution of [18F]JNJ-64511070 in Brain | Day 1
  The Distribution of [18F]JNJ-64511070 in brain will be measured by PET/CT scans obtained from the time of injection for up to 120 minutes along with measurement of the tracer input function with arterial samples for intact tracer and metabolites to establish the total and regional compartmental kinetics and volume of distribution (V[t]) of [18F]JNJ-64511070.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Approximately Up to 4 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Derived] Koole M, Schmidt ME, Hijzen A, Cohilis M, Vandermeulen C, Serdons K, Celen S, Bormans G, Maher M, Szardenings AK, Zhang W, Kolb H, de Hoon J, Van Laere K. Dosimetry and kinetic modelling of [18F]JNJ-64511070, a novel PET ligand to quantify AMPA-associated TARP-gamma8 receptors in the human brain. Eur J Nucl Med Mol Imaging. 2025 Dec;53(1):491-504. doi: 10.1007/s00259-025-07428-3. Epub 2025 Jul 22. PMID 40694102